CLINICAL TRIAL: NCT05775198
Title: Effects of Intrauterine Administration of Autologous Peripheral Blood Mononuclear Cells (PBMC) Immunomodulated With Interferon Tau (IFNt) Prior to Embryo Transfer on IVF Outcome
Brief Title: Effect of Intrauterine Administration of Autologous PBMC Modulated With IFNt on IVF Outcome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nadezhda Women's Health Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6/28022023
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Infertility, Female; IVF
Keywords: intrauterine PBMC; interferon tau; implantation; clinical pregnancy; live birth rate
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data analysis will be performed by investigators blind to the patient group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrauterine administration of PBMC immunomodulated with IFNt (Experimental): Approximately 9 ml whole blood will be collected from each patient 5 days post LH peak by peripheral venipuncture using a 21G butterfly catheter affixed via vacutainer to negative pressure receiving tubes (BD vacutainer acid-citrate-dextrose (ACD-A), REF:366645). PBMC will be isolated by density gradient centrifugation in room-temperature centrifuge set to 400 g for 25 min. After washing the obtained PBMCs, they will be suspended in RPMI 1640 supplemented with 10% HSA (human serum albumin) and incubated in the presence of 500 IU/ml IFNt for 24 h at 37˚C. On day 6 after LH peak, this cultured cell suspension will be carefully introduced in the uterine cavity by catheter. The following day (LH+7), patients will undergo a standard embryo transfer (ET) procedure.
  Interventions: Biological: PBMC immunomodulated with IFNt
- Control Group (No Intervention): Participants will undergo standard embryo transfer procedure with no intervention.

INTERVENTIONS:
Biological: PBMC immunomodulated with IFNt — Autologous peripheral blood mononuclear cells (PBMC) isolated using a standard protocol will be cultured in the presence of interferon tau (IFNt) for 24 hours at 37 ˚C and administered in the uterine cavity of patients 1 day prior to embryo transfer.
  Arms: Intrauterine administration of PBMC immunomodulated with IFNt

SUMMARY:
The goal of this clinical trial is to test the effect of modulated specialised immune cells isolated from the patients' own blood when administered to the uterus before embryo transfer on the IVF outcome (implantation, pregnancy and live birth rates).

To achieve this, blood will be obtained from eligible participants. Target cells will be isolated and incubated with the tested modulator for 24h, and returned to the uterine cavity 1 day prior to embryo transfer.

Researchers will compare the reproductive outcome of the tested intervention to that of a control group who will not receive the investigated cell treatment prior to embryo transfer.

DETAILED DESCRIPTION:
Female patients with no known uterine pathologies scheduled to undergo embryo transfer will be identified through patient records and invited to participate in the study. Five days after luteinizing hormone (LH) surge, peripheral blood mononuclear cells (PBMC) will be isolated from these patients' peripheral blood by density gradient centrifugation and suspended in culture medium. The obtained PBMC will be incubated with 500 IU/ml IFNt at 37˚C for 24 hours. This cell suspension will be carefully introduced in the uterine cavity by catheter on day 6 post LH surge. Embryo transfer will be performed the following day. A suitable age-matched control group will be recruited that will undergo embryo transfer but will not be administered immunomodulated PBMC prior to the transfer.

Reproductive outcomes in terms of rate of implantation, rate of clinical pregnancy and live birth rates will be recorded and compared between the two groups.

Data analysis will be performed by investigators blind to the patient group.

ELIGIBILITY:
Inclusion Criteria:

* Participating in Assisted Reproduction Treatment
* Having primary infertility
* Having regular menstrual cycles
* Scheduled to undergo embryo transfer of euploid embryos only

Exclusion Criteria:

* Uterine pathologies
* Endometrial bacterial infections
* Active endometrial inflammation
* Polycystic ovary syndrome
* Presence of auto antibodies such as anti-TPO (thyroid peroxidase), anti-TG (thyroglobulin), ACA (anticentromere antibodies), APA (antiphospholipid antibodies), ANA (antinuclear antibodies), and anti-dsDNA
* Presence of mutations involving the coagulation system such as deficiency of factor XII, Pro C, Pro S
* Oncological condition
* Positive HIV (human immunodeficiency virus), HCV (hepatitis C virus) or HBV (hepatitis B virus) tests

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-03-13 (Estimated); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
Rate of Implantation, % | 4 to 6 weeks post ET procedure
  Percentage of patients with positive hCG (human chorionic gonadotropin) test following ET
Clinical Pregnancy Rate, % | 6 weeks post ET procedure
  Percentage of patients with ultrasound confirmation of gestational sac or heartbeat following ET
Live Birth Rate, % | up to 10 months post ET procedure
  Percentage of patients with live birth following ET

CONTACTS AND LOCATIONS:
Locations (1):
- Nadezhda Women's Health Hospital, Sofia, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruseva M, Parvanov D, Ganeva R, Handzhiyska M, Safir J, Nikolova S, Tihomirova T, Metodiev D, Stamenov G, Hadjidekova S. Intrauterine Administration of PBMC Modulated with IFN-tau Before Embryo Transfer Improves Clinical Outcomes of IVF Patients-A Randomized Control Trial. Biomedicines. 2025 Dec 26;14(1):61. doi: 10.3390/biomedicines14010061. PMID 41595597